CLINICAL TRIAL: NCT07024238
Title: A Randomized Double Blinde Placebo-Controlled Trial of Short-Chain Fatty Acid Supplementation on Graft Function, Inflammatory Profile, and Microbiome Composition After Primary Kidney Transplantation
Brief Title: Impact of SCFA Supplementation on Gut Microbiome Composition of Kidney Transplant Recipients
Acronym: RENOBIOME
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Martin (Other)
Collaborators: Comenius University (Other)
Responsible Party: Principal Investigator, Matej Vnucak, deputy head of Transplant-nephrology Department, University Hospital, Martin
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TNO_UNM_SCFA2
Record Dates: First submitted 2025-04-22; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Effects; Immunosuppressive Agents; Renal Function; Adverse Events; Gut Microbiome; Flow Cytometry; Immune System; Metabolome
Keywords: short chain fatty acids; gut microbiome; kidney transplant recipients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCFA group (Experimental): Participants randomized at study with ID: TNO_UNM_SCFA1 to this group will receive 1000 mg of sodium butyrate daily for 12 weeks. The intervention aims to evaluate the effect of high-dose SCFA supplementation on the gut microbiome and systemic/urinary metabolome in kidney transplant recipients. The effect of different dosage of SCFA between study TNO_UNM_SCFA1 and TNO_UNM_SCFA2 will be examined also.
  Interventions: Dietary Supplement: SCFA
- Placebo group (Placebo Comparator): Participants in this group will receive placebo capsules identical in appearance to the active SCFA capsules, administered twice daily for 12 weeks. This arm serves as a control to evaluate the specific effects of SCFA supplementation.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: SCFA — Participants randomized to this group will receive 1000 mg of sodium butyrate daily for 12 weeks. The intervention aims to evaluate the effect of high-dose SCFA supplementation on the gut microbiome and systemic/urinary metabolome in kidney transplant recipients.
  Arms: SCFA group
Dietary Supplement: Placebo — Participants in this group will receive placebo capsules (sacharosis) identical in appearance to the active SCFA capsules, administered twice daily for 12 weeks. This arm serves as a control to evaluate the specific effects of SCFA supplementation.
  Arms: Placebo group

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the effects of high-dose short-chain fatty acid (SCFA) supplementation on the gut microbiome and host metabolome in stable kidney transplant recipients. Participants will be randomly assigned to receive either 1000 mg of sodium butyrate per day or placebo for a duration of 12 weeks. Comprehensive profiling of the serum and urinary metabolome, along with analysis of the gut microbiome composition and diversity, will be conducted at three time points: baseline, after the intervention period (week 12). The biochemical parameters and the level of tacrolimus will be also examined.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary kidney transplantation (living or dead donor)

Stable kidney transplant recipients (≥ 6 months post-transplantation)

Stable graft function defined as eGFR ≥ 30 mL/min/1.73 m² with no significant change (>15%) in the last 3 months

No episodes of acute rejection within the last 6 months

On stable immunosuppressive therapy for at least 3 months

Ability to provide written informed consent

Willingness and ability to provide stool, urine, and blood samples at specified time points

Exclusion Criteria:

* Use of antibiotics, probiotics, or prebiotics within 4 weeks prior to enrollment

Active gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, celiac disease)

Severe intestinal motility disorders or chronic diarrhea

Advanced liver disease (Child-Pugh C)

Active infection or systemic inflammatory disease requiring treatment

Uncontrolled diabetes mellitus (HbA1c > 9%)

Known allergy or intolerance to SCFA or ingredients in the supplement

Participation in another interventional clinical trial within the past 30 days

Pregnancy or breastfeeding

Hospitalization within 30 days prior to enrollment

Any condition which, in the opinion of the investigator, may compromise the safety of the participant or the integrity of the study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-09-04 (Estimated); Study Completion 2025-09-04 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiome composition after SCFA supplementation | Baseline to Week 12
  Evaluation of gut microbiota diversity and composition (alpha and beta diversity indices, relative abundance of microbial taxa) via 16S rRNA gene sequencing from stool samples.
Change in serum and urine metabolomic profile after higehr dose of SCFA supplementation | Baseline to Week 12
  Analysis of systemic metabolic changes using untargeted metabolomic profiling (NMR) in serum and urine samples and comarisation with results in study TNO_UNM_SCFA1.

SECONDARY OUTCOMES:
Safety and tolerability of high-dose SCFA supplementation | Baseline to Week 12
  Recording of adverse events (AEs), such as gastrointestinal symptoms.
Correlation between gut microbiome composition and serum metabolome. | Baseline to week 12
  Exploratory analysis of correlantion between gut microbiome composition and serum metabolites.
Intolerance of high dose SCFA. | Baseline to Week 12.
  Recording of treatment discontinuation rates due to intolerance or side effects.
correlantion between gut microbiome composition and urinary metabolites | Baseline to week12
  Exploratory analysis of correlantion between gut microbiome composition and urinary metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Martin, Martin, Slovakia, Slovakia

IPD SHARING:
Plan to Share IPD: No